CLINICAL TRIAL: NCT01421420
Title: Arizona Alzheimer's Disease Core Center
Brief Title: Alzheimer's Disease Core Center
Acronym: ADCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Arizona (Other)
Collaborators: Banner Health (Other); Barrow Neurological Foundation (Other); Mayo Clinic (Other); National Institute on Aging (NIA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: P30AG019610 (NIH); P30AG019610 (NIH)
Record Dates: First submitted 2011-07-25; First posted 2011-08-22 (Estimated); Last update posted 2015-06-12 (Estimated); Status verified 2015-01

CONDITIONS: Alzheimer's Disease; Mild Cognitive Impairment; Age-Related Memory Disorders
Keywords: Alzheimer's; Dementia; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction; Memory Disorders; Dementia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, brain tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Alzheimer's Disease
- Mild Cognitive Impairment
- Other forms of Dementia, not AD
- Normal Elderly Individuals

SUMMARY:
The main objective of this research project is to provide a comprehensive clinical database of patients with Alzheimer's disease (AD) and other forms of dementia, individuals with mild cognitive impairment (MCI), and age-matched normal controls. The study will also attempt to identify cognitively normal individuals at genetically defined risk for Alzheimer's disease through genetic screening.

All participants are seen annually. Autopsies to establish diagnoses in patients with dementia, patients with mild MCI, and cognitively normal elderly control subjects will also be conducted.

DETAILED DESCRIPTION:
All participants are seen annually. In addition to a detailed neurological examination, participants will receive a standardized battery of neuropsychological tests and will undergo genetic testing. The investigators will provide standardized periodic longitudinal assessment of the research participants. Autopsies to establish neurohistopathological diagnoses in clinically well-characterized patients with dementia, patients with mild MCI, and cognitively normal elderly control subjects will also be conducted.

ELIGIBILITY:
Inclusion Criteria:

For patients with MCI, or dementia, the presence of cognitive deficits including memory, language, and executive function.

Exclusion Criteria:

Presence of non-neurological medical conditions interfering with cognition.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Alzheimer's disease, mild cognitive impairment, other forms of dementia, and normal elderly individuals.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2001-07; Primary Completion 2024-12 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Neuropsychological Test Scores | Up to 20 years
  Cognitive function will be evaluated on a yearly basis using a battery of neuropsychological tests, which will then be scored and normed according to established guidelines.

SECONDARY OUTCOMES:
Neurological Exam | Up to 20 Years
  A thorough neurological exam will be performed once per year to evaluate neurological function.
Brain Tissue | From date of entry until date of death assessed up to 20 years
  A brain autopsy will be performed upon the participant's death to establish histological diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Z Rapcsak, M.D., Principal Investigator — University of Arizona
Locations (1):
- University of Arizona, University Medical Center, Tucson, Arizona, United States